CLINICAL TRIAL: NCT04030988
Title: The Reflection of Skin Color on the Efficacy of Narrow Band UVB in Stabilization of Active Cases of Vitiligo
Brief Title: Contribution of Skin Color in Stabilization of Active Cases of Vitiligo by Narrow Band UVB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Cairo University (Other); Menia University (Unknown); Suez Canal University (Other); Assiut University (Other); Alexandria University (Other)
Responsible Party: Principal Investigator, Mahy El-Bassiouny, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: u4xjkivz
Record Dates: First submitted 2019-04-22; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Vitiligo
Keywords: Vitiligo; Narrow-band UVB; Skin color; Minipulse
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: 100 patients with non-segmental vitiligo are randomized to either NB-UVB therapy with placebo versus NB-UVB combined with mini-oral pulse steroids therapy. Vitligo activity will be assessed according to the VIDA scoring system. Skin type, extent of vitiligo using VES score, photography of all areas according to the VES areas at a fixed distance of 50 cm from the patient, and using a 1 cm diameter circular white sticker for reference later will be done. All patients will receive NB-UVB phototherapy at starting dose of 0.3 J/cm2, 3 times per week for 6 months (72 sessions) with gradually increasing increments according until faint erythema is attained at which point the dose is fixed. 100 patients will be randomized into 2 groups; 50 patients will receive mini pulse dexamethasone therapy in a dose of 3 mg/ day for adults or 1.5 mg/day for children on two consecutive days per week while the other 50 patients will receive placebo having the same color, form and packaging for 6 months.
Who Masked: Care Provider
Masking Description: Masking involves only oral therapy; 100 patients will be randomized into 2 groups; 50 patients will receive mini pulse dexamethasone therapy in a dose of 3 mg/ day for adults or 1.5 mg/day for children on two consecutive days per week while the other 50 patients will receive placebo having the same color, form and packaging for 6 months.
  The investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): 50 patients will receive mini pulse dexamethasone therapy in a dose of 3 mg/ day for adults or 1.5 mg/day for children on two consecutive days per week plus NB-UVB phototherapy at starting dose of 0.3 J/cm2, at a rate of 3 times per week for 6 months (72 sessions) with gradually increasing increments.
  Interventions: Drug: Oral dexamethasone minipulse
- Placebo (Placebo Comparator): 50 patients will receive placebo having the same color, form and packaging as the dexamethasone therapy for 6 months plus NB-UVB phototherapy at starting dose of 0.3 J/cm2, at a rate of 3 times per week for 6 months (72 sessions) with gradually increasing increments.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Oral dexamethasone minipulse — 50 patients will receive mini pulse dexamethasone therapy in a dose of 3 mg/ day for adults or 1.5 mg/day for children on two consecutive days per week plus NB-UVB phototherapy at starting dose of 0.3 J/cm2, at a rate of 3 times per week for 6 months (72 sessions) with gradually increasing increments.
  Other Names: Narrow band UVB
  Arms: Active
Drug: Placebo oral tablet — 50 patients will receive placebo having the same color, form and packaging as the dexamethasone therapy for 6 months plus NB-UVB phototherapy at starting dose of 0.3 J/cm2, at a rate of 3 times per week for 6 months (72 sessions) with gradually increasing increments
  Other Names: Narrow band UVB
  Arms: Placebo

SUMMARY:
Vitiligo is a disease in which autoimmunity plays a major role. Multiple treatment options are available, of which narrow-band UVB is a cornerstone, acting through immunosuppression and repigmentation by stimulating reservoir melanocytes.

It's expected that this immunsupression is lower in darker skin types, where increased basal melanin might act as a barrier.

DETAILED DESCRIPTION:
Vitiligo is acquired depigmentation disorder. Several theories were hypothesized for causing vitiligo, of which the autoimmune theory is the most accepted.

The main targets of therapy are stabilization of the disease activity through immunosuppression, and repigmentation through stimulation of reservoir melanocytes proliferation and migration.

Narrow band ultraviolet phototherapy (NB-UVB) remains the cornerstone treatment of vitiligo. NB-UVB can induce both immunosuppression and repigmentation. Several factors can modulate the efficacy of NB-UVB therapy in treatment of vitiligo cases, including patient's age, lesion site, duration of the disease, and duration of the therapy.

The immunosuppressive function of NB-UVB was first detected in 1963 by Hanisko and Suskind, who observed that the contact hypersensitivity response in skin sensitized to dinitrochlorobenzene (DNCB) was reduced if skin was previously exposed to suberythemal doses of UVB.

Present evidence suggests that UVB suppress immune system through generation of T-suppressor cells, which inhibit the effector cells of Th1 type. It appears that UV-induced immunosuppression depresses the function of Th1 cells and enhances the activity of Th2 cells via cytokines such as Interleukin 10.

It's expected that this immunsupression is lower in darker skin types, where increased basal melanin might act as a barrier. However, skin was previously divided to UVB-resistant and UVB-sensitive (UVB-R and UVB-S) based on the contact hypersensitivity testing, regardless of the skin type. Moreover, A study on NB-UVB phototherapy for psoriasis revealed that photoadaptation during NB-UVB therapy Is Independent of skin type.

ELIGIBILITY:
Inclusion Criteria:

* Active cases of non-segmental vitiligo, VIDA +2 or more.
* All skin types
* Age above 6 years, both sexes.

Exclusion Criteria:

* Contraindications to NB-UVB ( photosensitive skin disorders, skin malignancy, patients on photosensitizing medications)
* Contraindications to mini-pulse steroid therapy (uncontrolled diabetes or hypertension, peptic ulcer)
* Stable disease (VIDA 0 & -1) and activity more than 6 months ago (VIDA +1).
* The use of other treatment for vitiligo during the 3 months previous to enrollment.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Detecting number of participants with clinical activity of vitiligo | At 6 months after treatment.
  Appearance of new lesions or expansion of pre-existing lesions by clinical examination.
Photography to detect activity of vitiligo | Change from baseline (first visit) at 6 months after treatment.
  New lesions in each area will be counted.
Elevation of serum Vitiligo activity markers. | Change from baseline at 6 months after treatment.
  A 5 cc blood sample will be withdrawn from each patient for:
  ELISA assessment of CXCL-10 (Pg/ml)
Elevation of PCR levels of serum Vitiligo activity markers | Change from baseline at 6 months after treatment.
  A 5 cc blood sample will be withdrawn from each patient for:
  PCR assessment of m-RNA of CXCL-10 as markers of disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mahy ElBassiouny, Ass.Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No
Methodology and outcome of the study is palnned to be published in an international medical journal with sharing participants data.